CLINICAL TRIAL: NCT02097979
Title: The Impact of a Brief Educational Intervention on Glaucoma Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Ellen Freeman, Associate Professor, Maisonneuve-Rosemont Hospital
Other Study IDs: Pfizer Canada NRA6110029
Record Dates: First submitted 2014-03-13; First posted 2014-03-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Glaucoma Medication Adherence
Keywords: glaucoma; adherence; medication possession ratio; intervention
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glaucoma Educational Intervention (Experimental)
  Interventions: Behavioral: Glaucoma Educational Intervention
- Delayed Intervention (No Intervention)

INTERVENTIONS:
Behavioral: Glaucoma Educational Intervention
  Arms: Glaucoma Educational Intervention

SUMMARY:
OBJECTIVE Our objective was to determine whether two group educational sessions plus one-on-one eye drop instillation training would improve adherence to glaucoma therapy as measured by pharmacy claims data in a cohort of newly diagnosed patients. Our hypothesis was that adherence would be improved in the intervention group and that patients would better understand their disease and how to manage it.

METHODS Study Design and Population: A randomized controlled clinical trial was conducted in newly diagnosed glaucoma patients at Maisonneuve-Rosemont Hospital in Montreal, Canada. Half of the participants were randomized to receive the intervention and half were randomized to receive a delayed intervention at the conclusion of the study. Inclusion criteria included a diagnosis of glaucoma requiring intraocular pressure lowering eye drop therapy and prescription drug insurance through the Régie de l'Assurance Maladie du Québec (RAMQ) (the Quebec Health Insurance Program) throughout the course of the study. There were three sources of data for this study: a questionnaire, the medical record, and RAMQ prescription drug claims data. Follow-up was for one year.

Recruitment and Randomization: From July, 2007 until December, 2011, a researcher approached eligible patients to determine their interest in participating in the study. Interested participants signed the informed consent form and were randomized. Participants in the intervention group were given an appointment to come back to the Hospital for the group intervention. Participants in the control group were given an appointment to receive the group intervention at the end of the study.

Intervention: Small groups of about 10 people were gathered for two 60-90 minute educational sessions on glaucoma in a classroom at Maisonneuve-Rosemont Hospital. During a break, each patient received one-on-one teaching on how to properly instill drops without touching the eye or using unnecessary drops.

Questionnaire and Assessment of Eye Drop Technique: A single questionnaire was given at the end of the study to all participants. The intervention group completed the questionnaire after the intervention while the control group completed the questionnaire before the intervention. Questions were included on demographics, systemic comorbidities, ocular medications, eye drop practices and difficulties, and glaucoma knowledge.

The instructor rated the ability of the participant to put eye drops in the eye taking into account the number of drops that were used and whether contact with the lid or conjunctiva occurred (good, fair, bad).

We created a composite score on the perception of the importance of glaucoma eye drop therapy using the following four questions: 1) do you think glaucoma is a serious disease, 2) do you believe that your treatment will be effective, 3) do you think your drops can lower the pressure in your eyes, 4) do you think your drops can help to preserve vision. Answers of no or do not know were given 0 points and answers of yes were given 1 point. Scores were summed and the composite score ranged from 0 to 4.

Medical Chart Review: At the end of the follow-up period, information was obtained on: the prescribed eye drop therapy for each patient per eye, whether the patient had undergone glaucoma filtering surgery, whether the patient had died or was no longer being followed, the most recent visual field mean deviation in the better eye using the Humphrey Visual Field Analyzer 24-2 SITA Standard Program.

Pharmaceutical Claims and Calculation of Medication Possession Ratio: The Medication Possession Ratio (MPR) was calculated as the sum of days of prescription supply divided by the number of days in which a prescription was required. Each person gave consent to contact the RAMQ to obtain pharmaceutical claims for all glaucoma medications. Data were collected on the date of purchase, and the name, dose, and class of the medicine. Data on the number of days of medication available per bottle were taken from the Rylander and Friedman studies with the minimum value used. For the numerator of the MPR, we calculated how many days of medication were available using RAMQ data. For the denominator of the MPR, we calculated the number of days that medication was prescribed in the medical chart. We took into account whether drops were needed for one or two eyes. If a participant was on multiple medications, we calculated a single mean MPR for all medications. We then dichotomized the MPR so that those having medication less than 75% of the days were defined as non-adherent, as we did previously in Djafari et al.

SIGNIFICANCE Adherence can be a problem in glaucoma because patients must often take daily eye drops despite not noticing any benefit to their vision and despite frequent side effects. Low cost interventions that help to improve adherence are needed.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria included a diagnosis of glaucoma requiring intraocular pressure lowering eye drop therapy and prescription drug insurance through the Régie de l'Assurance Maladie du Québec (the Quebec Health Insurance Program) throughout the course of the study.

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Medication Possession Ratio | 1-year post enrollment

SECONDARY OUTCOMES:
Eye drop instillation technique | At beginning or end of educational session
  Eye drop instillation technique was measured by direct observation. This was done in the experimental group immediately after the educational session and in the control group immediately before the educational session.
Perception of the importance of glaucoma eye drop therapy | At beginning or end of educational session
  Perception of the importance of glaucoma eye drop therapy was measured by questionnaire. In the experimental group this was done immediately after the educational session and in the control group this was done just before the educational session.

CONTACTS AND LOCATIONS:
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Djafari F, Lesk MR, Harasymowycz PJ, Desjardins D, Lachaine J. Determinants of adherence to glaucoma medical therapy in a long-term patient population. J Glaucoma. 2009 Mar;18(3):238-43. doi: 10.1097/IJG.0b013e3181815421. PMID 19295380